CLINICAL TRIAL: NCT04525677
Title: Gut Microbiome Dysbiosis in Sepsis-induced Coagulopathy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Zhi-jie He, Clinical Professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Other Study IDs: SYSEC-KY-KS-2020-107
Record Dates: First submitted 2020-08-20; First posted 2020-08-25 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In the diagnosis and treatment of patients with sepsis, through routine stool testing and dynamic testing of coagulation function, we found that patients often have stools that are not formed, the proportion of main fecal bacteria is imbalanced, the level of blood bacterial toxins rises, and the abnormal coagulation status indicate the gut microbiome dysbiosis may play an important regulatory role in abnormal blood coagulation in patients with sepsis. Therefore, we propose that the gut microbiome dysbiosis is involved in sepsis-induced coagulopathy. This project intends to prospectively observe the changes in gut microbiome dysbiosis and blood coagulation function in patients with sepsis before and after treatment, and explore whether the changes in gut microbiome dysbiosis promote the development of sepsis through coagulation disorders, provide new research perspectives for diagnosis and treatment for sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years and ≤85 years
* Sign the informed consent form
* Expected ICU hospital stay> 24 hours
* △SOFA score ≥2 and confirmed or suspected infection

Exclusion Criteria:

* Pregnant or breastfeeding women
* Estimated survival time <24 hours
* Diagnosis of sepsis time> 24 hours
* The length of ICU stay before diagnosis of sepsis> 7 days
* Sepsis from which the source of infection cannot be determined
* Congenital coagulopathy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Department of Intensive Care Unit, Sun Yat-sen Memorial Hospital, Sun Yat-sen University
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-07-15 (Actual); Primary Completion 2021-07-15 (Estimated); Study Completion 2021-07-15 (Estimated)

PRIMARY OUTCOMES:
Gut Microbiome alterations | Day 1- Day 14
  Taxonomic alterations,bacterial alpha diversity alterations,beta-diversity alterations of gut microbiome by performing metagenomic sequencing analysis of fecal samples
coagulation disorder tests | Day 1- Day 14
  Laboratory tests of coagulation disorder,such as PT,APTT,INR,TEG,fibrin degradation products , D-dimers.

CONTACTS AND LOCATIONS:
Overall Officials: minggen Zhou, Study Chair — Department of Intensive Care Unit, Sun Yat-sen Memorial Hospital, Sun Yat-sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China